CLINICAL TRIAL: NCT03511482
Title: An Open Feasibility Study to Investigate the Impact of A Digitally Delivered Asthma Service for Patients in Primary Care (IDEAL-001: Integrated Digitally EnhAnced Care for Long-term Conditions-001
Brief Title: Integrated Digitally Enhanced Care for Long-term Conditions- Asthma
Acronym: IDEAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: my mhealth Ltd (Industry)
Collaborators: Expert Health Ltd (Unknown); CLAHRC Wessex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IDEAL 001
Record Dates: First submitted 2018-04-04; First posted 2018-04-27 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Open Feasibility
Who Masked: Outcomes Assessor
Masking Description: The study will have a blinded team to perform final assesments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MyAsthma Application and Lloyds Pharmacy Online Doctor (Experimental): Web based applications to support people with Asthma management
  Interventions: Device: Lloyds Pharmacy Online Doctor
- MyAsthma Application and Usual care (Experimental): Web based application to support people with Asthma Management
  Interventions: Device: myAsthma Application
- Usual care only (control) (No Intervention): Usual care of asthma management

INTERVENTIONS:
Device: myAsthma Application — myAsthma Application is a Multi facetted online self management tool developed by my mhealth Ltd, which is an online interface for patient to feedback symptoms and (Quality of Life) QoL score. The app consists of an online action /self management plan, Patient education videos, medication diary, Peak Flow diary, Inhaler technique videos, mindfulness videos as well as weather and Pollution forecasters.
  Arms: MyAsthma Application and Usual care
Device: Lloyds Pharmacy Online Doctor — Online Doctor is part of Expert Health Ltd a doctor-led initiative providing safe and reliable remote online healthcare to adults in the UK. Their patient-centred model of healthcare allows patients to tailor care around their schedule and increases healthcare access for harder-to-reach patient groups.
  As the first ever online healthcare organisation to register with the government regulator of healthcare - and having received outstanding feedback from the Care Quality Commission about the high level of safe, effective, caring, responsive and well led care provided by the service - They pride themselves on their pioneer status and work constantly to expand the boundaries of personalised healthcare.
  Arms: MyAsthma Application and Lloyds Pharmacy Online Doctor

SUMMARY:
Asthma is a common lung condition that causes long term breathing difficulties. There is currently no cure for asthma but the use of simple inhaler treatments can keep the symptoms under control. If asthma symptoms get worse this can lead to an asthma attack which can be life-threatening. It has been shown that most of the deaths related to asthma are preventable if asthma is managed using the correct treatment plan however a significant proportion of patients are not using the right inhalers or not using them properly and do not know how to manage their asthma if it gets worse.

There is currently an unmet need to develop tools that can help improve asthma care, identify high risk patients, closely monitor their asthma control in 'real time' and intervene to optimise treatment to prevent asthma attacks. Both patients and indeed, the current British Thoracic Society (BTS) asthma guidelines recognise that technology has the potential to be used to improve asthma care and could lead to reductions in National Health Service (NHS) services use and improvements in symptoms.

Patients with better controlled asthma are less likely to be admitted to hospital and more likely to have an improved quality of life. This study aims to evaluate the delivery of an asthma service using an online doctor providing remote consultations paired with a self-management asthma app. The patients will use the app to input and track their symptoms, which will be monitored by a doctor remotely who can provide advice, optimise medications and intervene in a timely manner to prevent an asthma attack. The service is interactive, so the patient and doctor can communicate with one another 7 days a week by completing a consultation or sending messages via the online doctor portal or speaking on the telephone. The app will relay information about environmental triggers to the patient to help prevent the patient's asthma getting worse. The service will provide a new and potentially more convenient way of delivering routine appointments to reduce the numbers that do not attend. The patients will be able to watch educational videos stored on the app about asthma to potentially improve understanding of their condition. Digital training in inhaler technique will be supported with face to face support from pharmacists.

The goals are to increase adherence to and correct use of medication, help patients self-manage dynamically to reduce their risk of an asthma attack (with solutions personalised to an individual's triggers) and equip healthcare professionals with the data to identify those people at higher risk of an attack.

This is a before-and-after open interventional study, which means participants' asthma control will be compared before and after using the digital asthma management service. It is not a randomised study and participants will be given the choice of using a digital service. It is a single-centre study which will take place within one Clinical Commissioning Group (CCG) in Hampshire (UK), across at least two GP surgeries. It is anticipated that approximately 80 patients will be recruited.

Patients will be provided with this digital asthma service for a period of 6 months of 2018 and outcomes will be measured using a combination of questionnaires (quality of life, patient satisfaction, level of activation) and quantitative measures such as Forced Expired Volume over 1 second (FEV1)(measure of airway obstruction), Fractional Exhaled Nitric Oxide (FENO) (measure of airway inflammation) and Asthma Control Test Scores (measure of symptom control). Feedback from NHS professionals hosting the study and online doctors will also be sought. A Health economic model will be generated comparing the digitally enhanced model versus usual care. The main outcome of this study is looking at whether this new model of service delivery can provide an improvement in asthma control test scores.

DETAILED DESCRIPTION:
Asthma is a highly prevalent condition, which results from inflammation and hyper-responsiveness of the airways resulting in variable airway limitation and symptoms of wheeze, cough, breathlessness and chest tightness. 4.3 million adults (1 in 12) in the UK are currently receiving treatment for asthma. Treatment usually involves a combination of reliever and preventative inhaler therapy. On average 3 people a day die from asthma. The National Review of Asthma Deaths (NRAD) has shown that much of the morbidity relates to poor management particularly around the use of preventative treatment concluding that two-thirds of asthma deaths were preventable.

We have a well-established evidence base of how to help control asthma and prevent attacks using interventions that focus on maintaining control and reducing risk of an attack. However, there are concerns that the current National health Service (NHS) model of care: a once annual asthma review may not capture the full picture of asthma control and is generally limited to the period around that review, which is a fraction of the time people are living with asthma. Healthcare professionals aim to deliver the best care and motivate good asthma self-management, but this can be complex and time-consuming and so often is not possible in the allotted time for primary care appointments, leading to adverse outcomes and to variation in care.

Opportunities to address this variation in care were identified in the NRAD. These included improving risk stratification to distinguish between those with asthma requiring minimal support through an annual review and those who require closer monitoring throughout the year, ensuring safer prescribing to highlight where people with asthma have been prescribed excessive quantities of Short Acting Beta Agonist (SABA) inhalers, improving systems to arrange follow up, raising the quality of medical records and enabling systems to support asthma self-management.

The NHS spends around 1 billion a year treating and caring for people with asthma. Asthma accounts for about 60,000 hospital admissions per year. The annual 2016 asthma survey reported an overwhelming majority of patients, 82%, said their asthma was poorly controlled. Almost half of respondents said their asthma interfered with their day to day life and 46% said they had difficulty sleeping due to their asthma symptoms. Those with uncontrolled asthma were almost twice as likely to be admitted to hospital as those whose asthma symptoms were under control. The majority of patients admitted to hospital did not receive follow up putting them at higher risk of future attacks and re-admission to hospital. In the United Kingdom (UK) seven out of ten people with asthma receive care that fails to meet basic quality standards with 30-70% reported as not taking their asthma medication as prescribed.

With 85% of asthma patients being managed exclusively in primary care, asthma is estimated to account for around 2-3% of General Practitioners (GP) consultations19, costing an estimated £108 million annually. As highlighted by the recent General Practice Five Year Forward View, with an ever-increasing burden on services, conventional models of care are constantly being challenged and alternative, cost-effective ways of delivering healthcare to a larger cohort of patients are being sought.

Digital healthcare interventions may help to address some of these challenges by enabling remote delivery of patient-centred care, facilitating timely access to health advice and medications, prompting self-monitoring and medication compliance, and educating patients on trigger avoidance.

Telemonitoring, the transmission of monitoring data from a patient to an electronic health record which is shared with and monitored by healthcare professionals has the potential to improve outcomes. The impact of telemonitoring is likely to be strongly influenced by the level of professional support provided and personalisation of feedback. Studies have shown that people with poorly-controlled asthma have the potential to gain more by engaging with telemonitoring, helping people recognise worsening control and take preventative action to reduce their risk of an attack early. There is a substantial body of evidence to show that self-management education incorporating written personalised asthma action plans improves health outcomes for people with asthma. Self-management education reduces emergency use of healthcare resources including Accident and Emergency department visits and hospital admissions and improves markers of asthma control, including reduced symptoms and days off work and improved quality of life. Internet technology might offer an attractive means for encouraging patients to use self-management strategies within a day-to-day context.

In 2015, two thirds of patients with asthma had a smartphone, and with this ever-increasing presence of technology in homes, online prescribing and remote monitoring is beginning to emerge as an alternative way of delivering services. Nearly three-quarters of patients wanted to see an mHealth device that would help them monitor their asthma and nearly half would value a system which could be used as part of their asthma action plan and advise them if changes to medication have improved their asthma and when to seek medical attention. Three-quarters of healthcare professionals said they would value an mHealth system that would monitor patients' asthma symptoms over time and provide patients with an asthma action plan.

Systematic review has shown that despite the heterogenous interventions, technology enabled healthcare can improve process outcomes such as knowledge adherence to monitoring, self-management skills, improvement in inhaler technique and increased use of preventer medication. However, to date studies have shown an inconsistent effect on clinical outcomes such as symptoms lung function SABA use and quality of life. The use of computerised decision support systems need to align better with professional workflows so that pertinent and timely advice is easily accessible within the consultation. Evidence to support asynchronous remote consulting suggests that it leads to reductions in healthcare usage and disease status although evidence is very limited and of low quality in this patient group.

Systematic review of the use of technology enabled healthcare in asthma care has not identified significant harms or instances in which it was less effective than conventional care and the studies in asthma patients gave results encouraging enough to suggest further analysis of digital models of care. To the best of our knowledge, this is the first study looking at an integrated approach of using a self-management app, telemonitoring and asynchronous remote consulting in asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and over
* Able to give written informed consent
* A clinical diagnosis of Asthma on regular inhaled medication
* Measures of poor asthma control: Oral steroid use in the last 12 months and /or ACT score of less than 20 at screening, and/or use of 6 or more short acting beta-agonist inhalers in the last 6 months and/or frequent symptoms and/or (Accident and Emergency) A+E or hospital admission for asthma
* Access to the internet at home, use of mobile technology and the ability to operate a web platform in English
* No plans to travel abroad for prolonged periods during the trial period
* Consent to be contacted by phone, text and email

Exclusion Criteria:

* Asthma exacerbation in the past 4-6 weeks (Baseline visit to be delayed)

  . Patients who have a significant medical comorbidity that can present with asthma type symptoms e.g. COPD, Heart Failure, Lung Cancer (these cases require physical examination and a remote assessment would not be appropriate)
* Terminal Illness Pregnant
* Breast Feeding
* Patients who have another medical condition, including but not limited to respiratory immunological or cardiac disease other than asthma deemed by the investigators as significant
* Diagnosis of Occupational Asthma
* Patients on long term oral steroids or theophylline, as these treatments are not provided by the online doctor service
* Previous Intensive Therapy Unit (ITU) admission for asthma
* Patients under routine follow up of secondary care for asthmaHousebound
* Patients who are unable to read or use an internet-enabled device
* Alcohol and drug misuse
* Patients deemed unsuitable by their GP
* Patients who have another medical treatment(s), including but not limited to beta blockers deemed unsuitable by the investigators.

  * Already using a self management app.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-08 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | 12 months
  The ACT is a validated self administered questionnaire used to evaluate asthma control.ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning

SECONDARY OUTCOMES:
Incidence of treatment emergent Adverse and Serious Adverse Events (Safety and Tolerability | 12 months
  Safety assessed by the incidence of treatment pathway emergent adverse event (AE's) and Serious Adverse Events (SAE's) at study completion. The number of adverse events and serious adverse events will be tabulated also by the number patients reporting an event.
Patient Activation Measurement (PAM) | 12 months
  PAM is a tool used for measuring the level of patient engagement in their healthcare. It was designed to assess an individual's knowledge, skill and confidence for self-management. PAM is a 13-item scale that asks people about their beliefs, knowledge and confidence for engaging in a wide range of health behaviors and then assigns an activation score based on their responses to the 13-item scale. This will be assessed prior to and three months post intervention.
Asthma Exacerbation | 12 months
  Asthma exacerbation data will be collecting from their primary prescriber on their exacerbation history. The numbers of asthma exacerbations requiring oral antibiotics and/or oral steroids by the participants one year prior to starting the study will be recorded at visit one. If the participant has any exacerbations requiring oral antibiotics and/or steroids during the study period this will be recorded during monthly telephone contact with participants and at visit 2 .
Inhaler Technique | 12 months
  This will be assessed using the "7 Steps to successfully inhaler technique developed by the UK Inhaler Group. Each step is evaluated as being Good or Poor and the number of critical errors will be recorded.
Health Care Usage | 12 months
  Change in the median number of hospital and primary care interventions in the 6 months prior to the study and during the study period from baseline to study completion
Medication Adherence | 12 months
  Measure of primary and secondary medication adherence analysing prescription capture data, self-reported data via the MyAsthma app
Lung Function | 12 months
  Mean change in FEV1 from baseline to study completion - FEV1 will be obtained using spirometry. Spirometry will be performed at screening and end of study visit
Fractional Exhaled Nitric Oxide (FENO) | 12 months
  It is a simple breath test that measures the level of Nitric Oxide Concentration that the body naturally produces in the airways. FENo will be measured using a Bedfont device and will be performed at screening visit and end of study visit
Health Economics Analysis | 12 months
  The measurement of health outcome used will be the Quality Adjusted Life Year (QALY) calculated using the EQ5D-5L questionnaire.The EQ5D 5L is a validated questionnaire which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine.The use of NHS resources from an adjusted baseline period prior to staring the study compared to during the study will be used as a comparator for cost outcomes
Patient Health Questionnaire (PHQ9) | 12 month
  This is a self-administered validated questionnaire which scores each of the nine DSM-IV criteria as 0 (not at all) to 3 (nearly every day) and has been validated for use in primary care. It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment. Validity has been assessed against an independent structured mental health professional interview. PHQ-9 greater than or equal to 10 had a sensitivity of 88% and specificity of 88% for major depression. The questionnaire can be delivered over the telephone.
General Anxiety Disorder (GAD7) | 12 months
  The GAD-7 is a self-administered validated questionnaire and is used as a screening tool and severity measure for generalised anxiety disorder The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD. It is moderately good at screening three other common anxiety disorders - panic disorder (sensitivity 74%, specificity 81%), social anxiety disorder (sensitivity 72%, specificity 80%) and post-traumatic stress disorder (sensitivity 66%, specificity 81%).
Problematic Experiences of Therapy (PETS) | 12 months
  This is a validated questionnaire which measures difficulties experienced following the advice provided by an intervention.It has 4 domains which cover: 1) Whether symptoms themselves impede ability to follow advice, or are worsened by the advice, 2) Uncertainty about how to follow the advice, 3) Doubts about the efficacy of the app or online advice and 4) Practical obstacles to following the advice such as time or opportunity.
Self Efficacy for Appropriate Medication use Scale (SEAMS) | 12 months
  Was developed by a multidisciplinary team with expertise in medication adherence and health literacy. Its psychometric properties were then evaluated among 436 patients with coronary heart disease among other comorbid conditions. Reliability was evaluated by measuring internal consistency and test-retest reliability. The final 13 item scale showed good internal consistency reliability (Cronbach's alpha= 0.89). The SEAMS is a reliable and valid instrument that may provide a valuable assessment of medication self-efficacy in chronic disease management and appears to also be appropriate for use in patients with low literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Minal Bakhai, Principal Investigator — Lloyds Pharmacy Online Doctor
Locations (1):
- my mhealth Limited, Bournemouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Jong CC, Ros WJ, Schrijvers G. The effects on health behavior and health outcomes of Internet-based asynchronous communication between health providers and patients with a chronic condition: a systematic review. J Med Internet Res. 2014 Jan 16;16(1):e19. doi: 10.2196/jmir.3000. PMID 24434570
- [Background] Morrison D, Wyke S, Saunderson K, McConnachie A, Agur K, Chaudhuri R, Thomas M, Thomson NC, Yardley L, Mair FS. Findings from a pilot Randomised trial of an Asthma Internet Self-management Intervention (RAISIN). BMJ Open. 2016 May 12;6(5):e009254. doi: 10.1136/bmjopen-2015-009254. PMID 27173807
- [Background] Nystuen P, Hagen KB. Telephone reminders are effective in recruiting nonresponding patients to randomized controlled trials. J Clin Epidemiol. 2004 Aug;57(8):773-6. doi: 10.1016/j.jclinepi.2003.12.015. PMID 15485728
- [Background] Harris TJ, Carey IM, Victor CR, Adams R, Cook DG. Optimising recruitment into a study of physical activity in older people: a randomised controlled trial of different approaches. Age Ageing. 2008 Nov;37(6):659-65. doi: 10.1093/ageing/afn159. Epub 2008 Aug 20. PMID 18718924
- [Background] Treweek S, Pitkethly M, Cook J, Fraser C, Mitchell E, Sullivan F, Jackson C, Taskila TK, Gardner H. Strategies to improve recruitment to randomised trials. Cochrane Database Syst Rev. 2018 Feb 22;2(2):MR000013. doi: 10.1002/14651858.MR000013.pub6. PMID 29468635
- [Background] Leathem CS, Cupples ME, Byrne MC, O'Malley M, Houlihan A, Murphy AW, Smith SM. Identifying strategies to maximise recruitment and retention of practices and patients in a multicentre randomised controlled trial of an intervention to optimise secondary prevention for coronary heart disease in primary care. BMC Med Res Methodol. 2009 Jun 19;9:40. doi: 10.1186/1471-2288-9-40. PMID 19545366
- [Background] Braganza G, Chaudhuri R, McSharry C, Weir CJ, Donnelly I, Jolly L, Lafferty J, Lloyd SM, Spears M, Mair F, Thomson NC. Effects of short-term treatment with atorvastatin in smokers with asthma--a randomized controlled trial. BMC Pulm Med. 2011 Apr 7;11:16. doi: 10.1186/1471-2466-11-16. PMID 21473764
- [Background] Wright GR, Howieson S, McSharry C, McMahon AD, Chaudhuri R, Thompson J, Donnelly I, Brooks RG, Lawson A, Jolly L, McAlpine L, King EM, Chapman MD, Wood S, Thomson NC. Effect of improved home ventilation on asthma control and house dust mite allergen levels. Allergy. 2009 Nov;64(11):1671-80. doi: 10.1111/j.1398-9995.2009.02098.x. Epub 2009 Jul 24. PMID 19650848
- [Background] Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009 Oct;124(4):719-23.e1. doi: 10.1016/j.jaci.2009.06.053. Epub 2009 Sep 19. PMID 19767070
- [Background] Glaser, BG and Strauss, A. 1967. The discovery of grounded theory: Strategies for qualitative research, Chicago, IL: Aldine.
- [Background] Pope C, Mays N (2006) Qualitative Research in Health Care (3rd Edition) London: BMJ Books.
- [Background] Braun, V. and Clarke, V. (2006) Using thematic analysis in psychology. Qualitative Research in Psychology, 3 (2). pp. 77-101. ISSN 1478-0887 Available from: http://eprints.uwe.ac.uk/11735
- [Result] Bussey-Smith KL, Rossen RD. A systematic review of randomized control trials evaluating the effectiveness of interactive computerized asthma patient education programs. Ann Allergy Asthma Immunol. 2007 Jun;98(6):507-16; quiz 516, 566. doi: 10.1016/S1081-1206(10)60727-2. PMID 17601262
- [Result] Coffman JM, Cabana MD, Yelin EH. Do school-based asthma education programs improve self-management and health outcomes? Pediatrics. 2009 Aug;124(2):729-42. doi: 10.1542/peds.2008-2085. Epub 2009 Jul 27. PMID 19651589
- [Result] Guendelman S, Meade K, Benson M, Chen YQ, Samuels S. Improving asthma outcomes and self-management behaviors of inner-city children: a randomized trial of the Health Buddy interactive device and an asthma diary. Arch Pediatr Adolesc Med. 2002 Feb;156(2):114-20. doi: 10.1001/archpedi.156.2.114. PMID 11814370
- [Result] Bunting BA, Cranor CW. The Asheville Project: long-term clinical, humanistic, and economic outcomes of a community-based medication therapy management program for asthma. J Am Pharm Assoc (2003). 2006 Mar-Apr;46(2):133-47. doi: 10.1331/154434506776180658. PMID 16602223
- [Result] Hieftje K, Edelman EJ, Camenga DR, Fiellin LE. Electronic media-based health interventions promoting behavior change in youth: a systematic review. JAMA Pediatr. 2013 Jun;167(6):574-80. doi: 10.1001/jamapediatrics.2013.1095. PMID 23568703
- [Result] Pare G, Moqadem K, Pineau G, St-Hilaire C. Clinical effects of home telemonitoring in the context of diabetes, asthma, heart failure and hypertension: a systematic review. J Med Internet Res. 2010 Jun 16;12(2):e21. doi: 10.2196/jmir.1357. PMID 20554500
- [Result] Marcano Belisario JS, Huckvale K, Greenfield G, Car J, Gunn LH. Smartphone and tablet self management apps for asthma. Cochrane Database Syst Rev. 2013 Nov 27;2013(11):CD010013. doi: 10.1002/14651858.CD010013.pub2. PMID 24282112
- [Result] van der Meer V, Bakker MJ, van den Hout WB, Rabe KF, Sterk PJ, Kievit J, Assendelft WJ, Sont JK; SMASHING (Self-Management in Asthma Supported by Hospitals, ICT, Nurses and General Practitioners) Study Group. Internet-based self-management plus education compared with usual care in asthma: a randomized trial. Ann Intern Med. 2009 Jul 21;151(2):110-20. doi: 10.7326/0003-4819-151-2-200907210-00008. PMID 19620163
- [Result] de Jongh T, Gurol-Urganci I, Vodopivec-Jamsek V, Car J, Atun R. Mobile phone messaging for facilitating self-management of long-term illnesses. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007459. doi: 10.1002/14651858.CD007459.pub2. PMID 23235644
- [Result] DiBello K, Boyar K, Abrenica S, Worral PS. The effectiveness of text messaging programs on adherence to treatment regimens among adults aged 18 to 45 years diagnosed with asthma: a systematic review. JBI Database of Systematic Reviews and Implementation Reports 2014;12(1):485-532.
- [Result] Morrison D, Wyke S, Agur K, Cameron EJ, Docking RI, Mackenzie AM, McConnachie A, Raghuvir V, Thomson NC, Mair FS. Digital asthma self-management interventions: a systematic review. J Med Internet Res. 2014 Feb 18;16(2):e51. doi: 10.2196/jmir.2814. PMID 24550161
- [Result] Deshpande A, Khoja S, Lorca J, McKibbon A, Rizo C, Husereau D, Jadad AR. Asynchronous telehealth: a scoping review of analytic studies. Open Med. 2009 Jun 2;3(2):e69-91. PMID 19946396
- [Result] Matui P, Wyatt JC, Pinnock H, Sheikh A, McLean S. Computer decision support systems for asthma: a systematic review. NPJ Prim Care Respir Med. 2014 May 20;24:14005. doi: 10.1038/npjpcrm.2014.5. PMID 24841952
- [Result] Mukherjee M, Stoddart A, Gupta RP, Nwaru BI, Farr A, Heaven M, Fitzsimmons D, Bandyopadhyay A, Aftab C, Simpson CR, Lyons RA, Fischbacher C, Dibben C, Shields MD, Phillips CJ, Strachan DP, Davies GA, McKinstry B, Sheikh A. The epidemiology, healthcare and societal burden and costs of asthma in the UK and its member nations: analyses of standalone and linked national databases. BMC Med. 2016 Aug 29;14(1):113. doi: 10.1186/s12916-016-0657-8. PMID 27568881
- [Result] Ofcom, Communications Marketing Report (2015)
- [Result] Charlton I, White P. Asthma. Chapter 2.4. In: Jones R, Britten N, Culpepper L, Gass DA, Grol R, Mant D, et al. (eds). Oxford Textbook of Primary Medical Care, Vol. 2: clinical management. Oxford: Oxford University Press; 2004. pp. 682-90 20. Asthma UK. Annual Asthma Survey; 2016.
- [Result] Levy ML. National Review of Asthma Deaths (NRAD). Br J Gen Pract. 2014 Nov;64(628):564. doi: 10.3399/bjgp14X682237. No abstract available. PMID 25348975
- [Result] Car J, Sheikh A. Telephone consultations. BMJ. 2003 May 3;326(7396):966-9. doi: 10.1136/bmj.326.7396.966. No abstract available. PMID 12727771
- [Result] Car J, Sheikh A. Email consultations in health care: 2--acceptability and safe application. BMJ. 2004 Aug 21;329(7463):439-42. doi: 10.1136/bmj.329.7463.439. PMID 15321903
- [Result] McLean S, Sheikh A. Does telehealthcare offer a patient-centred way forward for the community-based management of long-term respiratory disease? Prim Care Respir J. 2009 Sep;18(3):125-6. doi: 10.3132/pcrj.2009.00006. No abstract available. PMID 19159046